CLINICAL TRIAL: NCT02037841
Title: The Impact of Implementing a Nursing-driven Clinical Pathway for Inpatient Management of Children Admitted to a Tertiary Care Centre With a Diagnosis of Asthma: A Randomized Controlled Trial
Brief Title: The Impact of Implementing a Nursing-driven Clinical Pathway for Inpatient Management of Children With Asthma
Acronym: NAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: CHAMO Innovation Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #11/10E
Record Dates: First submitted 2013-07-04; First posted 2014-01-16 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: Asthma; Nursing; Protocol; PRAM; Length of Stay; Weaning; Clinical pathway; Asthma exacerbation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nursing-driven Asthma protocol (Experimental): Children randomized to the intervention group will have their β2-agonist medication weaned by the nurse, according to the steps outlined in the clinical pathway. The nurse will ensure that the patient's family is booked for asthma teaching, and will also remind the physicians to fill out an asthma action plan on discharge. Detailed information as to when to contact physicians in the event of an acute deterioration of the patient is included in the clinical pathway.
  Interventions: Other: Nursing-driven clinical pathway for management of inpatient asthma
- Physician-driven asthma management (No Intervention): Patients in the control group will continue receiving the current standard of care, which consists of physicians weaning the β2-agonist medication when called to the bedside by the nurse or when deemed necessary by a physician

INTERVENTIONS:
Other: Nursing-driven clinical pathway for management of inpatient asthma
  Arms: Nursing-driven Asthma protocol

SUMMARY:
Asthma is the most common chronic disease of childhood and is responsible for large portion of pediatric admissions to Canadian hospitals. There is evidence that clinical pathways allow for optimal delivery of care and may result in decreased length of stay, leading to important economic benefits. Weaning of asthma medications prescribed for asthma exacerbation is not standardized in the current model of care. Currently, weaning is performed by ward physicians; in a teaching hospital, this most often done by residents staff. Differences in practice between different physicians, delays in patient assessment and adjustment of doctor's orders, likely prolong the hospital stay for children admitted with asthma.

This study's main objective is to determine the effect of a nursing-driven clinical pathway on children's length of stay when admitted to hospital with a diagnosis of acute asthma exacerbation. The pathway will allow nurses to wean a specific type of medication(β2-agonist), as compared to the current standard of care, which dictates that a physician writes an order to wean the medication. Number of administered β2-agonist treatments will be compared between both groups, as well as asthma-related health care utilization within two weeks of hospital discharge. Nursing, physician, and patients' satisfaction with the pathway will be evaluated, and a cost minimization analysis will be performed.

This study has the potential to improve resource use efficiency, increase patient safety by avoiding administration of unnecessary medications, and ameliorate quality of care by standardizing the care of children admitted to the hospital with a diagnosis of acute asthma exacerbation. The results of the study will be disseminated across the Canadian Health Care System with the goal of improving outcomes of children admitted to hospitals with acute asthma exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Children admitted during the study period with a diagnosis of asthma exacerbation, reactive airway disease, or wheezing
* Children aged 2 to 17 years

Exclusion Criteria:

* Children under the age of 2 years
* Children with congenital heart disease
* Children with chronic lung diseases other than asthma, including cystic fibrosis and bronchopulmonary dysplasia
* Children with severe neurological impairment
* Children with other significant co-morbid disorders
* Children whose caregivers do not understand English or French
* Children whose caregivers cannot be reached by phone for the 14-day follow up

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2012-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Length of hospital admission, in hours | Duration of hospital admission, average 2-3 days
  The participants will be followed for the duration of their hostpital admission, an expected average of 2-3 days.

SECONDARY OUTCOMES:
The number of inhaled or nebulized β2-agonist treatments given | Duration of hospital admission, average 2 -3 days
  The participants will be followed for the duration of their hostpital admission, an expected average of 2-3 days.
number of children transferred to the ICU | During admission to hospital, average 2-3 days
  The participants will be followed for the duration of their hostpital admission, an expected average of 2-3 days.
number of families attending asthma teaching sessions | Duration of hospital admission, average 2-3 days
  The participants will be followed for the duration of their hostpital admission, an expected average of 2-3 days.
number of children seeking medical attention for asthma-related issues | Within 2 weeks of hospital discharge date
  Follow up will occur to assess all children who seeked medical attention for concerns related to asthma for two weeks post-discharge from hospital
Nursing and physician satisfaction with the pathway | At study completion, expected within 2 to 3 years
patient satisfaction with the care received in hospital | Within 2 weeks of hospital discharge date
  Follow up satisfaction questionaire will be completed within two weeks of discharge from hospital

OTHER OUTCOMES:
Cost analysis | At study completion, expected within 2-3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada